CLINICAL TRIAL: NCT01067118
Title: Ultra-Short Acting Insulin Versus Short Acting Insulin Effect on Postprandial Hyperglycemia AKA RCT Comparing Linjeta Versus Humalog in Pumps: Effect on Postprandial Glycemia
Brief Title: A Randomized Control Trial Comparing Linjeta Versus Humalog in Pumps: Effect on Postprandial Blood Sugars.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was suspended due to lack of study drug
Sponsor: Stanford University (Other)
Collaborators: Biodel (Industry); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Bruce A. Buckingham, Principle Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: SU-01292010-4823; 17579
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Humalog U-100 Insulin (Active Comparator)
  Interventions: Drug: Humalog U-100
- LINjeta U-100 (Experimental)
  Interventions: Drug: LINjeta U-100 Insulin

INTERVENTIONS:
Drug: LINjeta U-100 Insulin — LINjeta U-100 Insulin will be used per the subjects normal insulin carbohydrate and insulin sensitivity factors
  Other Names: VIAject U-100
  Arms: LINjeta U-100
Drug: Humalog U-100 — Normal short acting insulin used in participants daily life including carbohydrate ratios and insulin sensitivity factors
  Other Names: Lispro U-100 insulin
  Arms: Humalog U-100 Insulin

SUMMARY:
The purpose of this study is to determine if the use of Linjeta(tm) insulin when compared to Humalog will result in significantly lower episodes of hyperglycemia and hypoglycemia after a breakfast meal.

ELIGIBILITY:
Inclusion Criteria:1)Type 1 diabetes for at least 1 year

1. The diagnosis of type 1 diabetes is based on the investigator¡-s judgment; C peptide level and antibody determinations are not needed.

   2) Age : 18 years old ¨C 49.99 years old 3) Continuous subcutaneous insulin infusion (CSII) therapy for at least 3 months 4) Participant consent demonstrated by signing IRB approved documents 6) HgA1c ¡Ü 9% 7) If participant is female with reproductive potential, willing to avoid pregnancy and pregnancy test negative. Exclusion Criteria:1) Chronic oral steroid use

   2) The presence of a significant medical disorder that in the judgment of the investigator will affect the wearing of sensors or the completion of any aspect of the protocol.

   3) Known clinical history of celiac disease or inflammatory bowel disease. 4) Participants will have a negative anti-endomysial antibody or anti-tissue transglutaminase antibody within one year of enrollment.

   5) Cystic Fibrosis 6) Inpatient psychiatric treatment in the past 6 months. 7) Currently pregnant or lactating, or anticipate getting pregnant in the next one year.

   8) Clinical diagnosis of gastroparesis. 9) Insulin binding capacity greater than 10 microunits per litter

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint for this first phase is the 3 hour area under the curve from baseline following a standardized breakfast meal. | 2 weeks
The primary endpoint for this second phase is the 3 hour area under the curve from baseline following a standardized breakfast meal in the outpatient setting. | 2 weeks
The primary endpoint for this third phase is daytime (6 am to midnight) average glucose values.is percent of CGMS glucose values in range (70-180 mg/dL) for the third week fo sensor data in each group. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A. Buckingham, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado Denver School of Medicine Barbara Davis Center, Denver, Colorado